CLINICAL TRIAL: NCT03507751
Title: Pharmacokinetics of Meropenem During High-dose Continuous Renal Replacement Therapy in Critically Ill Patients
Brief Title: Pharmacokinetics of Meropenem During High-dose CRRT
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Collaborators: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Michał Borys, M.D., Ph.D., Medical University of Lublin
Other Study IDs: 90/2009/IV
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Infection; Renal Failure
MeSH Terms: conditions — Infections; Renal Insufficiency | interventions — Meropenem

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for obtaining meropenem concentrations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Meropenem: Patients who require meropenem and CRRT during ICU (intensive care unit) stay
  Interventions: Drug: Meropenem; Device: CRRT

INTERVENTIONS:
Drug: Meropenem — 1.0 gram of meropenem given intravenously every 8 hours
Device: CRRT — Continuous renal replacement therapy for three days

SUMMARY:
Assessment of meropenem plasma concentration in critically ill patients who require CRRT (continuous renal replacement therapy). A standard dose of meropenem is administered, i.e. 1 gram every 8 hours.

DETAILED DESCRIPTION:
This is a prospective observational study performed on critically ill patients. Inclusion criteria are a severe infection on admission requiring the use of meropenem and CRRT.

Both medical and surgical patients will be included. Any type of infections can be included (pulmonary, abdominal, urinary tract, etc.) Antibiotics regimen includes one-hour infusion of meropenem (1.0 gram) intravenously every 8 hours.

Blood samples (2 mL) will be collected at the 15, 30, 45, 60, 75, 90, 120, 180, 240, and 480 minutes after each dose of meropenem for 3 consecutive days. The standard arterial canula will be used to obtain samples.

30 minutes after each sample collection, blood will be centrifuged for 10 minutes at 3,000 rpms. Subsequently, supernatant will be collected and frozen.

Serum meropenem concentration will be measured by high-performance liquid chromatography.

Each patient's hemodynamic parameters will be recorded with the use of transpulmonary thermodilution technique (PICCO). Other therapies, i.e. ventilatory support, sedation, an antifungal agent will be given as required.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require ICU treatment due to severe infection
* age 18-80 years
* an eligible consent obtained from the patient or his/her attendant

Exclusion Criteria:

* allergy to meropenem
* lack of consent to participate in the study
* age of patients below 18 or above 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely ill patients treated in ICU
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of meropenem | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Oddział Kliniczny Anestezjologii i Intensywnej Terapii, Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No